CLINICAL TRIAL: NCT06844188
Title: The Effect of Prenatal Education at Pregnancy School on Primary Cesarean Rate
Brief Title: The Effect of Prenatal Education on Primary Cesarean Rate
Status: Completed | Type: Observational
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SEAH_birth
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-02

CONDITIONS: Prenatal Care Late; Cesarean Delivery Affecting Fetus
Keywords: prenatal care; cesarean section; prenatal education; primary cesarean

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective case-control study examining the impact of antenatal education on mode of delivery. The study will include all deliveries occurring between January 2024 and December 2024. Participants will be divided into two groups: a case group consisting of women who attended antenatal classes (pregnancy school) and a control group of women who did not. The primary outcome will be mode of delivery (vaginal or cesarean).

The study will collect data on gravida and parity. Participants will be further categorized into four groups based on their delivery history:

Women undergoing a cesarean section for their first delivery. Women experiencing a normal vaginal delivery for their first delivery. Women with a history of vaginal delivery who have another vaginal delivery in this pregnancy.

Women with a history of vaginal delivery who deliver via cesarean section in this pregnancy.

Each of these four groups will have a corresponding case (antenatal class attendees) and control (non-attendees) subgroup.

Data on cesarean section indications, the name of the physician performing the cesarean, and the hospital's annual primary cesarean section rates will be requested from the hospital and compared across groups. For the case group, information regarding the specific antenatal education received, the gestational week at which the education was received, and patient characteristics such as age, infant birth weight, and educational level will also be collected.

DETAILED DESCRIPTION:
Inclusion Criteria:

All women who gave birth between January 2024 and December 2024 and attended antenatal classes (pregnancy school) will be included in the study.

For the control group (women who did not attend antenatal classes), participants will be randomly selected, matching the case group (antenatal class attendees) in terms of age, education level, and parity.

Exclusion Criteria:

Women with a history of previous cesarean sections who are undergoing a repeat cesarean in this pregnancy will be excluded.

Women with high-risk pregnancies, such as preeclampsia, preterm labor, preterm premature rupture of membranes, multiple pregnancies, previous cesarean section, or placental abruption, will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

All women who gave birth between January 2024 and December 2024 and attended antenatal classes (gebe okulu) will be included in the study.

For the control group (women who did not attend antenatal classes), participants will be randomly selected, matching the case group (antenatal class attendees) in terms of age, education level, and parity.

Exclusion Criteria:

Women with a history of previous cesarean sections who are undergoing a repeat cesarean in this pregnancy will be excluded.

Women with high-risk pregnancies, such as preeclampsia, preterm labor, preterm premature rupture of membranes, multiple pregnancies, previous cesarean section, or placental abruption, will not be included in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant
Study Population: pregnant women of prenatal educated and prenatal non-educated about birth
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
primary cesarean rate | 1 year
  rates of cesarean

CONTACTS AND LOCATIONS:
Overall Officials: Alev esercan, M.D., Study Director — Sanliurfa Education and Research Hospital
Locations (1):
- Sanliurfa Training and Resarch Hospital, Sanliurfa, Turkey (Türkiye)